CLINICAL TRIAL: NCT03029026
Title: A sTudy invesTigating the Role of Occult cArdiaC Amyloid in The Elderly With Aortic Stenosis
Brief Title: The Role of Occult Cardiac Amyloid in the Elderly With Aortic Stenosis.
Acronym: ATTRact-AS
Status: Completed | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 006974
Record Dates: First submitted 2017-01-09; First posted 2017-01-24 (Estimated); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Amyloidosis; Aortic Stenosis
Keywords: Cardiac amyloidosis; Aortic stenosis; DPD scintigraphy
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Aortic Valve Stenosis | interventions — Caves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples will be biobanked for all patients (n=250). Endomyocardial biopsy specimens will be snap frozen and biobanked for those patients undergoing sAVR (n=50).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Those patients for TAVR: Those patients who are undergoing TAVR (clinical decision) who are recruited at the Barts Heart Centre will undergo clinical echocardiography, research DPD scintigraphy and clinical TAVR work-up CT (with research post contrast acquisitions at 3-5 minutes), unless already performed prior to recruitment. Those patients undergoing TAVR (clinical decision) who are recruited at the John Radcliffe Hospital will undergo clinical echocardiography and research DPD scintigraphy only. N=150.
  Interventions: Other: Baseline assessment; Procedure: Transthoracic echocardiography; Procedure: 99mTc-3,3-diphosphono-1,2-propanodicarboxylic acid scintigraphy; Radiation: CT 3-5-minute post-contrast research sequences; Other: Follow-up assessment
- Those patients for sAVR: Those patients who are undergoing sAVR (clinical decision) will undergo clinical echocardiography, research DPD scintigraphy, research CMR and endomyocardial biopsy at the time of surgery. N=50.
  Interventions: Other: Baseline assessment; Procedure: Transthoracic echocardiography; Procedure: 99mTc-3,3-diphosphono-1,2-propanodicarboxylic acid scintigraphy; Procedure: Cardiac Magnetic Resonance; Procedure: Endomyocardial biopsy; Other: Follow-up assessment
- Those patients for medical management: Those patients who are decided for medical management (clinical decision) will undergo clinical echocardiography, research DPD scintigraphy and any other imaging as per work-up/trial prior to no intervention decision. N=50.
  Interventions: Other: Baseline assessment; Procedure: Transthoracic echocardiography; Procedure: 99mTc-3,3-diphosphono-1,2-propanodicarboxylic acid scintigraphy; Other: Follow-up assessment

INTERVENTIONS:
Other: Baseline assessment — Baseline assessment will include clinical history, Quality of Life Questionnaire (EQ-5D/SF-12), a 6-minute-walk test, blood sampling for haematocrit, renal function, biomarkers (NT-pro-BNP and troponin), and biobanking (also for AL exclusions if scanning positive), a urine sample for biobanking (also for AL exclusions if scanning positive), as well as tests performed as the routine pre-operative work-up (clinical electrocardiogram, blood pressure to estimate global LV afterload, valvulo-arterial impedance).
Procedure: Transthoracic echocardiography — Patients will undergo a clinical transthoracic echocardiogram for the assessment of AS severity and diastolic function in line with the British Society of Echocardiography guidance. Simultaneous, optimised 2-chamber, 3-chamber and 4-chamber views will need to be recorded (over 3 cycles) for strain analysis.
  Severe AS will be defined using standard echocardiography guidelines in conjunction with MDT consensus.
  Other Names: Echo
Procedure: 99mTc-3,3-diphosphono-1,2-propanodicarboxylic acid scintigraphy — Scanning will use a hybrid SPECT-CT gamma camera after intravenous injection of 700 MBq of DPD (effective dose 4mSv). Acquisition technique: 5-minute (early) and then 3-hour (late) whole body planar scans, followed by SPECT-CT of the heart. Qualitative visual (Perugini) scoring of the cardiac uptake is performed from the 3-hour whole body planar images and the SPECT-CT images.
  Other Names: DPD scintigraphy
Radiation: CT 3-5-minute post-contrast research sequences — Cardiac CT for ECV will use the dedicated cardiac CT scanner (Somatom FORCE; Siemens Medical Solutions, Germany). 3-5-minute post contrast research images will be taken at the end of the clinically indicated TAVR work-up CT.
  Other Names: ECV by CT
  Groups: Those patients for TAVR
Procedure: Cardiac Magnetic Resonance — CMR will be performed using a 1.5-T Aera for standard late gadolinium enhancement, as well as T1 mapping and ECV.
  Other Names: CMR
  Groups: Those patients for sAVR
Procedure: Endomyocardial biopsy — Septal tissue specimens will be taken under direct vision by the surgical team using a 14-gauge coaxial needle system. Biopsies will be screened for amyloid by Congo red staining; if positive, tissue will be fully sub-typed (immunohistochemistry, mass spectrometry).
  Groups: Those patients for sAVR
Other: Follow-up assessment — 1-year follow-up with clinical echocardiogram (for sAVR and TAVI patients) and/or telephone interview for all patients (if not carried out in person at the time of the echocardiogram). This will include a follow up Quality of Life Questionnaire as per baseline. If attending clinic or echocardiogram a 6-minute-walk test will also be performed.

SUMMARY:
Aortic stenosis (AS) is the most common valvular heart disease. Once symptomatic with severe AS, outcome is poor unless the valve is replaced surgically or via transcatheter aortic valve replacement (TAVR). Transthyretin amyloid (ATTR) deposits are common in the heart muscle in up to 25% of octogenarians, and after an asymptomatic period of unknown duration, cause overt heart failure and arrhythmias in a proportion of cases. The prevalence and impact of covert ATTR amyloidosis in elderly individuals with AS are unknown. Detection would avoid misdiagnosis, guide treatment and, potentially, improve outcomes. Recent data have shown that echocardiography, cardiovascular magnetic resonance (CMR), computed tomography (CT), and DPD scintigraphy, can identify ATTR amyloid deposits, but the clinical performance of these various tests is unknown.

This study will investigate elderly patients with symptomatic severe AS using imaging to explore ATTR amyloid in AS and determine its prevalence and impact on outcome.

The investigators aim to recruit a total of 250 patients aged 75 or older being considered for intervention for severe AS. The prevalence of cardiac amyloid will be assessed in three arms (sAVR, TAVI and medical therapy, with a likely patient ratio of 50:150:50), using five investigation modalities - all cohorts (echocardiography and DPD scintigraphy); sAVR cohort (biopsy and CMR); TAVI cohort (EqCT); medical therapy only cohort (as per work-up/trial prior to no intervention decision).

The primary outcome measure is patient mortality. Secondary outcomes measures are major adverse cardiovascular events, length of stay, pacemaker implantation, ECV measured by EqCT and CMR.

Follow up will be at 1-year with clinical echocardiogram (for sAVR and TAVI patients) and/or telephone interview for all patients (if not carried out in person at the time of the echocardiogram).

DETAILED DESCRIPTION:
INTRODUCTION

Calcific aortic stenosis (AS) is the most common valve disease in the West with a prevalence of 2.8% in patients over 75 years. Once symptomatic with severe AS, outcome is poor, unless the valve is replaced surgically (sAVR) or via transcatheter aortic valve replacement (TAVR), which is predominantly used in elderly patients for whom surgery is deemed too high risk.

Systemic amyloidosis is a multisystem disease characterised by extracellular deposition of abnormally folded protein, which over time results in progressive organ dysfunction. These protein deposits bind Congo red stain, producing the pathognomonic apple-green birefringence under polarised light. Cardiac involvement is the leading cause of morbidity and mortality in these patients. Amyloidosis due to transthyretin deposition (ATTR) can be due to wild-type transthyretin amyloid deposits, also known as senile systemic amyloidosis, which predominantly accumulates in the heart. Primary light chain (AL) amyloidosis and hereditary transthyretin amyloidosis can also affect the heart.

Wild-type ATTR (wtATTR) amyloid deposition is present in up to a 25% of individuals aged over 85 at autopsy. To date, this has been no more than an academic observation, but technology is changing this: cardiac imaging, particularly cardiovascular magnetic resonance (CMR) and 99mTc-3,3-diphosphono-1,2-propanodicarboxylic acid (DPD) scintigraphy, can now detect the disease antemortem, which is generating a major increase in national awareness. There are also significant advances being made in the treatment of amyloidosis. There are several drugs in clinical trial including novel antisense and interfering RNA therapeutics that can reduce production of TTR by up to 80-90%. Also on the horizon are treatments to promote clearance of established amyloid, notably including monoclonal anti-SAP (serum amyloid P component) antibodies. Despite the prevalence of wtATTR amyloid deposits at autopsy, their clinical significance and prognostic impact of in severe AS has not been explored.

Co-existent cardiac amyloid and AS. Given the prevalence of wtATTR in octogenarians at autopsy, AS and wtATTR are likely to co-exist - the literature has early evidence for this. In a cohort of 20 patients with AS, who had undergone TAVI and subsequently valve explantation at autopsy (n=17) or surgery (n=3), cardiac amyloid was found in a third of these patients and was thought to contribute to death in the majority. Our research also supports this - the "RELIEF-AS" study. In 146 patients with severe AS undergoing sAVR, we found cardiac amyloid deposits in 6 patients. All were wtATTR, all calcific AS, with the youngest patient being aged 69. Comprehensive imaging was performed, which showed a diagnostic imaging hierarchy: echocardiography was non-contributory, CMR detected a third of cases, whereas DPD scintigraphy was positive in all four patients scanned (2 died before the test). Biopsy ATTR deposits were prognostic and the strongest predictor of adverse outcome - regardless of infiltration degree or its imaging detection: post sAVR 50% with wtATTR died by 1 year vs 9% without (p<0.001). Occult amyloid has also been implicated in the need for pacemakers in TAVR patients.

The availability of TAVI has extended the range of individuals that can benefit from intervention for AS, prolonging life. TAVR patients are generally older so more likely to have wtATTR. One recent abstract found a 16% (23% in men) prevalence of cardiac amyloid in in patients undergoing TAVR (n=75) using 99mTc-pyrophosphate scintigraphy (PYP, a bone tracer available in the USA, which is possibly inferior to DPD). WtATTR is also an increasingly recognized cause of heart failure with preserved ejection fraction (HFpEF). DPD scintigraphy in 120 hospitalized patients who also had LV wall thickness ≥12 mm and an EF ≥50%, showed that 16 patients (13.3%) showed moderate to severe myocardial uptake.

Why detect wtTTR amyloid in severe AS? There are two separate aspects of wtATTR in AS. First, wtATTR in patients with moderate AS may mimic severe AS, (particularly low-flow, low-gradient) causing misdiagnosis. Second, wtATTR may itself be a disease modifier, leading to a more severe phenotype with more heart failure, arrhythmia, and higher mortality. We think there is a large, now detectable, UK population of elderly patients undergoing sAVR or TAVR with a significant occult amyloid. This could influence therapeutic options (TAVR vs sAVR vs medical therapy), intervention timing and medications - specific amyloid therapies, drugs to avoid (e.g. digoxin and diltiazem).

How to detect wtATTR? There are multiple techniques that could detect cardiac wtATTR. Each has their pros and cons with different evidence bases. Our initial study used three imaging modalities and biopsy to detect the presence of cardiac amyloid in sAVR. DPD scintigraphy was the superior imaging modality, with the highest diagnostic sensitivity. There is now a rapidly growing body of evidence supporting DPD scintigraphy as the non-invasive investigation of choice for diagnosing cardiac ATTR. A recent multi-centre study of over 1,000 patients showed that bone scintigraphy had a >99% sensitivity for cardiac ATTR deposits and they proposed it should have a role in diagnosing the condition without the need for invasive cardiac biopsy, which has previously been considered the gold standard.

The investigators have recently created a new modality: equilibrium contrast computed tomography (EqCT), which requires a single extra image dataset of the heart to be taken 5 minutes after the routine TAVR work-up CT images are taken. Extracellular volume fraction (ECV) calculated by EqCT discriminated 100% between cardiac amyloid involvement and patients with AS in 53 patients.

TRIAL OBJECTIVES

Hypothesis:

In the elderly with severe AS being considered for intervention (TAVR, sAVR), wtATTR is:

* Common.
* Conveys a worse prognosis.
* Can be reliably detected non-invasively.

Aim:

To confirm the prevalence, clinical impact (procedural complications, symptom response to aortic valve replacement, 1-year mortality) and potential place of imaging (DPD scintigraphy, ECV by CT, CMR and echocardiography) in occult amyloid in severe AS.

STUDY PLAN

Design: prospective observational cohort with 1 year follow-up.

Population: patients aged 75 or older with severe AS referred to the Barts Heart Centre for consideration for intervention (sAVR or TAVR) or referred to the John Radcliffe Hospital in Oxford for consideration for TAVR.

Proposed sample size: two centre study (Barts Heart Centre and the John Radcliffe Hospital), 250 patients.

Recruitment: patients will be recruited from General Cardiology, TAVR and Cardiothoracic Surgery Outpatient Clinics. A large proportion of these patients are discussed in the Valve Multidisciplinary Team Meeting, which will provide another source of recruitment. This will take place over an 18-month period from August 2016 to February 2018.

Baseline assessment: will include clinical history, Quality of Life Questionnaire (EQ-5D/SF-12), a 6-minute-walk test, blood sampling for haematocrit, renal function, biomarkers (NT-pro-BNP and troponin), and biobanking (also for AL exclusions if scanning positive), a urine sample for biobanking (also for AL exclusion if scanning positive), as well as tests performed as the routine pre-operative work-up (clinical electrocardiogram, blood pressure to estimate global LV afterload, valvulo-arterial impedance).

Measures of exposure: the prevalence of cardiac amyloid assessed in three arms (sAVR, TAVI and medical therapy, with a likely patient ratio of 50:150:50), using five investigation modalities - all cohorts (echocardiography and DPD scintigraphy); sAVR cohort (biopsy and CMR); TAVR cohort (EqCT); medical therapy only cohort (as per work-up/trial prior to no intervention decision).

Follow-up: 1-year follow-up with clinical echocardiogram (for sAVR and TAVR patients) and/or telephone interview for all patients (if not carried out in person at the time of the echocardiogram). This will include a follow up Quality of Life Questionnaire as per baseline. If attending clinic or echocardiogram a 6-minute-walk test will also be performed. MACE and mortality endpoints will also be identified.

ELIGIBILITY:
Inclusion Criteria:

* Aged 75 or above
* Severe aortic stenosis being considered for intervention
* Patient informed consent

Exclusion Criteria:

* Unable to provide informed consent
* Patient declined or withdrew consent (at any stage)
* Imaging modality specific contraindications:

  1. Being considered for sAVR, however unsuitable for study CMR due to contraindications such as a device in situ, severe claustrophobia, renal impairment (eGFR <30) or previous severe gadolinium contrast allergy.
  2. Being considered for TAVR work-up CT, however unsuitable for contrast due to previous severe iodinated contrast allergy. NB patients with significant renal impairment are given pre-hydration routinely by the managing clinicians.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with symptomatic severe AS being considered for intervention.
Sampling Method: Non-Probability Sample
Enrollment: 581 (Actual)
Dates: Start 2011-02-22 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Patient mortality | Through study completion, an average of 1 year
  From patient notes, GP records or Office of National Statistics.

SECONDARY OUTCOMES:
Major adverse cardiovascular events (MACE) | Post-TAVI investigation - 1-year
  From patient's medical records. Includes for example: cardiac death, myocardial infarction and emergency cardiac surgery or intervention.
Length of hospital stay | Post-TAVI investigation - 1-year
  From patient's medical records
Pacemaker implantation | Post-TAVI investigation - 1-year
  From patient's medical records
Outcome of the various cardiac imaging modalities | 1-year
  From patient's medical records

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Barts Heart Centre, London
  - The John Radcliffe Hospital, Oxford

REFERENCES:
- [Background] Lindroos M, Kupari M, Heikkila J, Tilvis R. Prevalence of aortic valve abnormalities in the elderly: an echocardiographic study of a random population sample. J Am Coll Cardiol. 1993 Apr;21(5):1220-5. doi: 10.1016/0735-1097(93)90249-z. PMID 8459080
- [Background] Kvidal P, Bergstrom R, Horte LG, Stahle E. Observed and relative survival after aortic valve replacement. J Am Coll Cardiol. 2000 Mar 1;35(3):747-56. doi: 10.1016/s0735-1097(99)00584-7. PMID 10716479
- [Background] Banypersad SM, Moon JC, Whelan C, Hawkins PN, Wechalekar AD. Updates in cardiac amyloidosis: a review. J Am Heart Assoc. 2012 Apr;1(2):e000364. doi: 10.1161/JAHA.111.000364. Epub 2012 Apr 24. No abstract available. PMID 23130126
- [Background] Falk RH. Diagnosis and management of the cardiac amyloidoses. Circulation. 2005 Sep 27;112(13):2047-60. doi: 10.1161/CIRCULATIONAHA.104.489187. No abstract available. PMID 16186440
- [Background] Tanskanen M, Peuralinna T, Polvikoski T, Notkola IL, Sulkava R, Hardy J, Singleton A, Kiuru-Enari S, Paetau A, Tienari PJ, Myllykangas L. Senile systemic amyloidosis affects 25% of the very aged and associates with genetic variation in alpha2-macroglobulin and tau: a population-based autopsy study. Ann Med. 2008;40(3):232-9. doi: 10.1080/07853890701842988. PMID 18382889
- [Background] Coelho T, Adams D, Silva A, Lozeron P, Hawkins PN, Mant T, Perez J, Chiesa J, Warrington S, Tranter E, Munisamy M, Falzone R, Harrop J, Cehelsky J, Bettencourt BR, Geissler M, Butler JS, Sehgal A, Meyers RE, Chen Q, Borland T, Hutabarat RM, Clausen VA, Alvarez R, Fitzgerald K, Gamba-Vitalo C, Nochur SV, Vaishnaw AK, Sah DW, Gollob JA, Suhr OB. Safety and efficacy of RNAi therapy for transthyretin amyloidosis. N Engl J Med. 2013 Aug 29;369(9):819-29. doi: 10.1056/NEJMoa1208760. PMID 23984729
- [Background] Ackermann EJ, Guo S, Booten S, Alvarado L, Benson M, Hughes S, Monia BP. Clinical development of an antisense therapy for the treatment of transthyretin-associated polyneuropathy. Amyloid. 2012 Jun;19 Suppl 1:43-4. doi: 10.3109/13506129.2012.673140. Epub 2012 Apr 12. PMID 22494066
- [Background] Richards DB, Cookson LM, Berges AC, Barton SV, Lane T, Ritter JM, Fontana M, Moon JC, Pinzani M, Gillmore JD, Hawkins PN, Pepys MB. Therapeutic Clearance of Amyloid by Antibodies to Serum Amyloid P Component. N Engl J Med. 2015 Sep 17;373(12):1106-14. doi: 10.1056/NEJMoa1504942. Epub 2015 Jul 15. PMID 26176329
- [Background] Nietlispach F, Webb JG, Ye J, Cheung A, Lichtenstein SV, Carere RG, Gurvitch R, Thompson CR, Ostry AJ, Matzke L, Allard MF. Pathology of transcatheter valve therapy. JACC Cardiovasc Interv. 2012 May;5(5):582-590. doi: 10.1016/j.jcin.2012.03.012. PMID 22625199
- [Background] Kim WK, Rolf A, Liebetrau C, Van Linden A, Blumenstein J, Kempfert J, Bachmann G, Nef H, Hamm C, Walther T, Mollmann H. Detection of myocardial injury by CMR after transcatheter aortic valve replacement. J Am Coll Cardiol. 2014 Jul 29;64(4):349-57. doi: 10.1016/j.jacc.2014.03.052. PMID 25060368
- [Background] Castano A, Bokhari S, Maurer MS. Could late enhancement and need for permanent pacemaker implantation in patients undergoing TAVR be explained by undiagnosed transthyretin cardiac amyloidosis? J Am Coll Cardiol. 2015 Jan 27;65(3):311-2. doi: 10.1016/j.jacc.2014.09.084. No abstract available. PMID 25614433
- [Background] Gonzalez-Lopez E, Gallego-Delgado M, Guzzo-Merello G, de Haro-Del Moral FJ, Cobo-Marcos M, Robles C, Bornstein B, Salas C, Lara-Pezzi E, Alonso-Pulpon L, Garcia-Pavia P. Wild-type transthyretin amyloidosis as a cause of heart failure with preserved ejection fraction. Eur Heart J. 2015 Oct 7;36(38):2585-94. doi: 10.1093/eurheartj/ehv338. Epub 2015 Jul 28. PMID 26224076
- [Background] Gillmore JD, Maurer MS, Falk RH, Merlini G, Damy T, Dispenzieri A, Wechalekar AD, Berk JL, Quarta CC, Grogan M, Lachmann HJ, Bokhari S, Castano A, Dorbala S, Johnson GB, Glaudemans AW, Rezk T, Fontana M, Palladini G, Milani P, Guidalotti PL, Flatman K, Lane T, Vonberg FW, Whelan CJ, Moon JC, Ruberg FL, Miller EJ, Hutt DF, Hazenberg BP, Rapezzi C, Hawkins PN. Nonbiopsy Diagnosis of Cardiac Transthyretin Amyloidosis. Circulation. 2016 Jun 14;133(24):2404-12. doi: 10.1161/CIRCULATIONAHA.116.021612. Epub 2016 Apr 22. PMID 27143678
- [Background] Treibel TA, Bandula S, Fontana M, White SK, Gilbertson JA, Herrey AS, Gillmore JD, Punwani S, Hawkins PN, Taylor SA, Moon JC. Extracellular volume quantification by dynamic equilibrium cardiac computed tomography in cardiac amyloidosis. J Cardiovasc Comput Tomogr. 2015 Nov-Dec;9(6):585-92. doi: 10.1016/j.jcct.2015.07.001. Epub 2015 Jul 10. PMID 26209459
- [Background] Perugini E, Guidalotti PL, Salvi F, Cooke RM, Pettinato C, Riva L, Leone O, Farsad M, Ciliberti P, Bacchi-Reggiani L, Fallani F, Branzi A, Rapezzi C. Noninvasive etiologic diagnosis of cardiac amyloidosis using 99mTc-3,3-diphosphono-1,2-propanodicarboxylic acid scintigraphy. J Am Coll Cardiol. 2005 Sep 20;46(6):1076-84. doi: 10.1016/j.jacc.2005.05.073. PMID 16168294
- [Derived] Smith A, Fullerton J, Whittle J, Moon J, Mullen M, Scully P, Hamilton-Davies C. Relationship between endotoxin core and staphylococcal antibody levels and outcome following transcatheter aortic valve implantation (TAVI). Perioper Med (Lond). 2025 Aug 14;14(1):87. doi: 10.1186/s13741-024-00464-x. PMID 40813990
- [Derived] Patel KP, Scully PR, Saberwal B, Sinha A, Yap-Sanderson JJL, Cheasty E, Mullen M, Menezes LJ, Moon JC, Pugliese F, Klotz E, Treibel TA. Regional Distribution of Extracellular Volume Quantified by Cardiac CT in Aortic Stenosis: Insights Into Disease Mechanisms and Impact on Outcomes. Circ Cardiovasc Imaging. 2024 May;17(5):e015996. doi: 10.1161/CIRCIMAGING.123.015996. Epub 2024 May 21. PMID 38771906
- [Derived] Scully PR, Patel KP, Klotz E, Augusto JB, Thornton GD, Saberwal B, Haberland U, Kennon S, Ozkor M, Mullen M, Lloyd G, Kelion A, Menezes LJ, Hawkins PN, Moon JC, Pugliese F, Treibel TA. Myocardial Fibrosis Quantified by Cardiac CT Predicts Outcome in Severe Aortic Stenosis After Transcatheter Intervention. JACC Cardiovasc Imaging. 2022 Mar;15(3):542-544. doi: 10.1016/j.jcmg.2021.10.016. Epub 2021 Dec 15. No abstract available. PMID 34922871
- [Derived] Scully PR, Treibel TA, Fontana M, Lloyd G, Mullen M, Pugliese F, Hartman N, Hawkins PN, Menezes LJ, Moon JC. Prevalence of Cardiac Amyloidosis in Patients Referred for Transcatheter Aortic Valve Replacement. J Am Coll Cardiol. 2018 Jan 30;71(4):463-464. doi: 10.1016/j.jacc.2017.11.037. No abstract available. PMID 29389364